CLINICAL TRIAL: NCT04814784
Title: Retrospective Study Comparing Neoadjuvent Short Course of Radiotherapy to Conventional Chemoradiation in Cancer Rectum
Brief Title: Role of Neoadjuvent Radiotherapy in Locally Advanced Cancer Rectum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amany sayed Abass (Other)
Responsible Party: Sponsor-Investigator, Amany sayed Abass, Physician Dr, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Radiotherapy in rectal cancer
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Neoadjuvent radiotherapy either short or long course chemoradiation in treatment of locally advanced cancer rectum — Study the effect of neoadjuvent radiotherapy in treatment of locally advanced cancer rectum e higher possiblity of preservation of anal sphincter and decreased rate of locoregional recurrence compared to surgery alone

SUMMARY:
This is a retrospective study comparing neoadjuvent short course radiotherapy to conventional chemoradiation in locally advanced cancer rectum and the effect of both regimens in overall survival and disease free survival

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer diagnosed in the western world. In 2019 there were approximately 44180 new cases of rectal cancer diagnosed in the United states.

Due to the close proximity of the rectum to pelvic structures and organs, the absence of a serious membrane surrounding the rectum and the restriction of the surgical view and access by the pelvic cavity, the locoregional recurrence rate in rectal cancer is relatively high after surgery alone.

Neoadjuvent therapy rather than surgery followed by adjuvent therap has been the preferred approach world wide in treatment of rectal cancer since the 2004 publication of the seminal German CAO/ARO/AIO-94 study ,which compared preoperative with postoperative chemoradiation in 823 patients The use of neoadjuvent therapy is recommended for all newly diagnosed rectal adenocarcinoma with a clinical stage T3 or T4 based on trans rectal endoscopic ultrasound or pelvic MRI .Neoadjuvent therapy may comprise of either radiotherapy alone or in combination with chemotherapy, commonly prescribed chemotherapy agents include 5-fluorouracil and Oxaloplatin.

Both short course radiotherapy (25 Gy in 5 fractions) and long course radiotherapy (50.4Gy in 28 fractions, conventionally fractionated therapy)can be applied as neoadjuvent radiotherapy.

Several phase lll RCTs,including three large well-designed international RCTs have reported that short course neoadjuvent radiation treatment improves local control compared with surgery alone in patients with respectable rectal cancer.

Also ,neoadjuvent chemoradiation with long course radiotherapy can be recommended for most patients with stage ll- lll rectal cancer with the aim of reducing the risk of local recurrence, for reducing rates of perioperative and post operative complications and in an attempt to avoid radical surgery with permanent colostomy.

ELIGIBILITY:
Inclusion Criteria:

* histologically proved adenocarcinoma of the rectum
* Age between 18 and 70 yrs
* T3 and T4 N1,N2 respectable tumor
* The WHO performance score 0-2
* have a free metastatic work up excluded by chest x-ray , abdominal ultrasonography or CT pelviabdomen

Exclusion Criteria:

* patients with locally advanced inoperable disease locally recurrent rectal cancer
* had a history of malignant tumor within 5 years except the skin cancer
* pregnant or lactating women
* previous irradiation in pelvis
* there was contraindication for neoadjuvent radiotherapy or surgery
* known metastatic disease
* mental disorder

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Locally advanced cancer rectum patients stage ll ,lll who received neoadjuvent radiotherapy either short or long course chemoradiation before surgery
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Effect of neoadjuvent radiotherapy in treatment of locally advanced cancer rectum | 4 years
  Disease free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt cancer Institute, Asyut, Egypt

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Song JH, Jeong JU, Lee JH, Kim SH, Cho HM, Um JW, Jang HS; Korean Clinical Practice Guideline for Colon and Rectal Cancer Committee. Preoperative chemoradiotherapy versus postoperative chemoradiotherapy for stage II-III resectable rectal cancer: a meta-analysis of randomized controlled trials. Radiat Oncol J. 2017 Sep;35(3):198-207. doi: 10.3857/roj.2017.00059. Epub 2017 Sep 15. PMID 29037017
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Rodel C, Liersch T, Becker H, Fietkau R, Hohenberger W, Hothorn T, Graeven U, Arnold D, Lang-Welzenbach M, Raab HR, Sulberg H, Wittekind C, Potapov S, Staib L, Hess C, Weigang-Kohler K, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R; German Rectal Cancer Study Group. Preoperative chemoradiotherapy and postoperative chemotherapy with fluorouracil and oxaliplatin versus fluorouracil alone in locally advanced rectal cancer: initial results of the German CAO/ARO/AIO-04 randomised phase 3 trial. Lancet Oncol. 2012 Jul;13(7):679-87. doi: 10.1016/S1470-2045(12)70187-0. Epub 2012 May 23. PMID 22627104
- [Background] Li Y, Wang J, Ma X, Tan L, Yan Y, Xue C, Hui B, Liu R, Ma H, Ren J. A Review of Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer. Int J Biol Sci. 2016 Jul 17;12(8):1022-31. doi: 10.7150/ijbs.15438. eCollection 2016. PMID 27489505